CLINICAL TRIAL: NCT06794632
Title: A Protocol for a Randomised Controlled Pilot and Feasibility Study
Brief Title: Cross-sectorial Management Program for People Living with Hand Osteoarthritis: a Randomised Controlled Pilot and Feasibility Study
Acronym: HANDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Research Institute (Other)
Responsible Party: Principal Investigator, Eva Ejlersen Wæhrens, Professor, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HANDY pilot-RCT
Record Dates: First submitted 2025-01-07; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hand Osteoarthritis
Keywords: Hand osteoarthritis; Activity of Daily Living; Group intervention

STUDY DESIGN:
Intervention Model Description: The study is designed as a two-armed parallel pilot RCT following the CONSORT guideline - extension for pilot and feasibility trials. Following baseline assessments, participants will be randomised either to the HANDY occupational therapy intervention or usual care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HANDY occupational therapy intervention (Experimental): Group-based occupational therapy
  Interventions: Other: HANDY occupational therapy intervention
- Waiting list (No Intervention): Waiting list will receive no intervention (usual care)

INTERVENTIONS:
Other: HANDY occupational therapy intervention — The HANDY occupational therapy intervention is occupation-centred and follows the Occupational Therapy Intervention Process Model (OTIPM), specifying the steps of a problem-solving process focused on enabling performance of tasks in everyday life. The HANDY occupational therapy intervention consists of six mandatory sessions of 120 minutes representing a combination of individual and group sessions. Each group includes a maximum of eight participants with hand osteoarthritis, facilitated by two OTs.
  Arms: HANDY occupational therapy intervention

SUMMARY:
To investigate the research design (pilot-RCT) and feasibility of the HANDY program for people with hand osteoarthritis (version 2.0). In collaboration with two municipalities (Lyngby-Taarbæk and Ballerup), the research design is tested in a pilot-RCT before planning a full-scale RCT study. The entire HANDY program is described in a manual, which has been adjusted to version 2.0 based on a previous feasibility study. The focus of the study will be on procedures related to recruitment and retention, the study's acceptance in practice, and the appropriateness of assessment tools in connection with the occupational therapy group intervention. The feasibility and acceptance of the HANDY program version 2.0 are also examined in this study.

DETAILED DESCRIPTION:
Background Globally, nearly 600 million people are affected by osteoarthritis (OA), causing pain and stiffness (1). Hand OA (HOA) is the second most common subtype of OA. People with HOA often experience decreased ability to perform Activities of Daily Living (ADL) (2,3)This includes Personal ADL (PADL) tasks such as getting dressed, eating, and performing manicure, and Instrumental ADL (IADL) tasks, such as hot and cold meal preparation, cleaning, and bicycling (4). Research suggests that occupational therapy interventions are effective in improving ADL ability among people with chronic conditions (5-7). Still, rigorous studies, testing the outcomes of occupational therapy introducing compensatory strategies (e.g., strategy training, assistive devices, and splints) to reduce symptoms and improve ADL ability in people with HOA are limited (8,9). Furthermore, a recent audit among Danish general practitioners (n=348) indicates that among people with HOA experiencing decreased ADL ability (n=147) only one was referred for occupation therapy (10).

Accordingly, to ensure that people with HOA are referred for and will receive effective occupational therapy interventions, the development of a multidisciplinary cross-sectorial management program for people with HOA, named HANDY, was initiated in 2023. In the development process, the United Kingdom's Medical Research Council's (MRC) framework for developing and evaluating complex interventions was employed (11). The MRC framework prescribes four phases: 1) development, 2) feasibility/piloting, 3) evaluation, and 4) implementation (11). As recommended by the MRC framework, a core element in the development of the HANDY program has been the involvement of stakeholders through co-productional activities (12) to ensure the sustainability of the HANDY program. Accordingly, the content and delivery of the HANDY program was based on the experiences and preferences among people with HOA, clinicians (i.e., general practitioners (GPs), occupational therapists (OTs), rheumatologists), and previous research (5,13-18).

The manualised HANDY program consists of two parts: an organizational part and an occupational therapy intervention part. The organizational part includes 1) a needs evaluation conducted by the GP to clarify the client's need for referral to occupational therapy, 2) procedures for referral for occupational therapy in the municipality, and 3) procedures for the cross-sectorial communication and collaboration between the GP and OT (19). The occupational therapy part of the program will be delivered in the municipality and includes: an individual session evaluating the ADL ability of the person with HOA and establishing goals for the intervention; four group-based sessions involving peer-learning activities using compensatory strategies; homework between sessions; and an individual session re-evaluating the individual's ADL ability(19).

A feasibility study, of the first version of the HANDY program (v1.0), based on the guidance developed by O'Cathain and al (20), was carried out from January to June 2024, addressing the following feasibility aspects (19): 1) Intervention development, 2) Intervention components, 3) Perceived value, benefits, harms or unintended consequences, 4) Acceptability in principle, 5) Feasibility and acceptability in practice, and 6) Fidelity, reach and dose. The results of the feasibility study revealed needs to i) improve identification of people with HOA in need for occupational therapy in the general practices; ii) establish a stronger connection between the evaluation of ADL ability and goal setting (first session) and the solutions presented in the group sessions; iii) improve the learning activity designed to support participants in gaining a transactional understanding of their problems with ADL, and iv) improve procedures for homework. Based on these results, the second version of the HANDY program (v2.0) was developed.

In accordance with the MRC framework (11) and the guidelines by O'Cathain and al. (20), the next step will be to conduct a study to evaluate remaining feasibility aspects and pilot aspects of trial design, conduct and processes, outcomes, and measures, prior to initiating a full scale randomised controlled trial (RCT) of the HANDY program (v.2.0).

Methods Specific aims

Based on the guidance by O'Cathain and al. (20), the specific study aims are to:

1. Pilot central aspects of trial design, conduct and processes in terms of:

   * effectiveness of recruitment, randomisation, and retention (Recruitment and retention).
   * acceptability of study procedures (Acceptability of the trial in practice).
   * appropriateness of outcomes and measurements (Breadth and selection of outcomes)
   * completion of outcome measures (Completion of measures)
2. Evaluate remaining feasibility aspects:

   * Explore mechanisms of actions assumed to be essential for the HANDY occupational therapy intervention to produce the intended outcomes (Mechanisms of action).
   * Explore if the revised HANDY program (v 2.0) is feasible and acceptable, based on adjustments made (Feasibility and acceptability in practice).

Study design and settings The HANDY pilot study is designed as a two-armed parallel RCT following the CONSORT guideline (21). Following baseline assessments, participants will be randomised either to the HANDY occupational therapy intervention or usual care. Since people with HOA rarely are referred from GP to OT, usual care represents no intervention. Accordingly, to mimic real-life settings and enhance the applicability of the study results, the control group will consist of a waiting list. Outcomes assessments will be carried out at baseline and post intervention (week 7). After study completion, participants in the control group will be offered the occupational therapy intervention part of the HANDY program.

The study will be conducted between January 1st and June 30th, 2025, in two municipalities previously involved in the feasibility study of the HANDY 1.0 program, both located in the Capital Region of Denmark (19).

Participants and recruitment People diagnosed by GP with HOA, aged > 18 years, experiencing decreased ADL ability due to HOA, without severe vision and hearing loss, or cognitive deficits affecting the ability to engage in peer-learning activities and group discussions. People unable to participate in two or more group sessions due to other scheduled activities (e.g. holidays/travels) are not eligible. Furthermore, people where acute illness is the primary reason for decreased ADL ability, will be referred to other services in the municipality.

Participants with HOA will be recruited through various approaches. First, GPs working in general practices in the municipalities involved will be introduced to the needs evaluation and referral procedures of the HANDY program (v2.0) and asked to suggest study participation to people in their clinic with need for occupational therapy due to HOA. Second, posters informing on the HANDY pilot study will be posted in GP clinics and municipal rehabilitation centres. The posters will include information about who will be eligible, study period, and encourage people with HOA experiencing decreased ADL ability to ask their GP for a referral. Also, contact information to researchers will be provided, if any question arises or the need of assistance occurs.

The GP will decide if referral for occupational therapy is relevant, based on the needs evaluation. When the referral for occupational therapy is received in the municipality, the person with HOA meeting the study inclusion criteria will be informed about the pilot study and invited to participate. Information will include allocation, trial procedures, and the rights to withdraw. If the person wants to participate in the study, written consent is obtained. People not meeting the inclusion criteria or not interested in study participation, will be offered a standard occupational therapy session to clarify if other municipal services are relevant.

OTs, working in each of the municipal rehabilitation centres involved, with at least six months of working experience in this type of setting will be responsible for the delivery of the HANDY program. To support the delivery, the OTs will be trained in procedures related to the HANDY program v2.0.

The HANDY program Organisational part (Needs evaluation, referral and communication) The needs evaluation is conducted by the GP to determine if the HOA affects the client's performance of ADL tasks. It is based on the GP's assessment and the client's perspective. First, the GP asks questions on how the person with HOA perceives using the hands in performance of ADL tasks (e.g., zipping zippers when dressing, cutting nails, opening cans when cooking, or wringing a cloth when cleaning). Then a screening involving seven aspects is conducted: 1) decreased grip strength, 2) problems turning things with the hands, for example turning a key in a lock, or turning a rounded doorknob or handle, 3) problems related to turning taps on and off, 4) problems peeling vegetables or fruit, 5) problems picking up big, heavy thing, 6) problems wringing a washcloth or dishcloth, and 7), problems related to buttoning buttons. Grip strength is assessed using simple handshake (i.e., GP's assessment), and the remaining aspects are assessed by asking the person with HOA (i.e., self-report). All aspects are rated as "yes" or "no". The person with HOA is referred to occupational therapy based on rating at least one of the five aspects as "yes".

Referral is conducted using existing electronic procedures. As part of the referral the GP takes an anamnesis focusing on the level of functioning and the identified problems related to ADL. Also, the specific diagnosis is included. In the municipality, the referral is received and processed according to standard procedures.

Immediately after the final session of the occupational therapy intervention, the OT submits a medical discharge summary to the GP, representing the primary part of the cross-sectorial communication and Collaboration. The summary includes information on the level of goal-attainment, obtained changes in ADL-I and AMPS measures, descriptions of any referrals to other services (e.g., assistive devices or assistance in the home) and future recommendations.

Occupational Therapy Intervention The HANDY occupational therapy intervention is occupation-centred and follows the Occupational Therapy Intervention Process Model (OTIPM) (22), specifying the steps of a problem-solving process focused on enabling performance of tasks in everyday life. The HANDY occupational therapy intervention consists of six mandatory sessions of 120 minutes representing a combination of individual and group sessions. Each group includes a maximum of eight participants with HOA, facilitated by two OTs.

Session 1 consists of an individual session in the person with HOA's home involving evaluations of self-reported and observed ADL task performance. The Activities of Daily Living Interview (ADL-I) is used to measure self-reported ADL ability (23), and the Assessment of Motor and Process Skills (AMPS) to measure observed ADL ability (24,25). Both ADL-I and AMPS are valid and reliable measurements for people with chronic conditions. Following the ADL evaluations, the person with HOA and the OT will together formulate goals for the intervention using the Goal Attainment Scale (GAS) (26) and together consider reasons for decreased ADL ability.

Sessions 2 to 5 are group-based, held at the rehabilitation centre, and involve peer learning activities. In session 2 the people with HOA are introduced to how a transactional perspective can identify factors not only related to hand function but influencing their individual ADL task performances (22). The results of the individual analyses form the basis for sessions 3 to 5 focusing on improving ADL task performance by addressing these factors. The HANDY occupational therapy intervention is mainly based on compensatory strategies to improve ADL task, in relation to energy conservation (session 3), assistive devices and the use of orthoses (session 4). The last group sessions (session 5) will also address how a broader spectrum of tasks (e.g., ADL, leisure, or social activities) may be used to maintain hand function. The group sessions will be individualised based on the people with HOA's individual evaluations and problems performing ADL tasks. The HANDY occupational therapy intervention is terminated with an individual session (session 6) in the person with HOA's home involving evaluation of goal attainment and changes in self-reported and observed ADL ability using ADL-I, AMPS and GAS (23-26).

Program theory As recommended by the MRC framework (11), a preliminary program theory has been developed, describing how the program is expected to lead to its outcomes and in what circumstances. The program theory addresses four aspects of the program: an occupation-centred paradigm, supportive institutional contexts, the need for systematic evaluations, and group peer-exchange as a mean to facilitate change.

Based on the results of the feasibility study (19), three specific topics in the preliminary program theory will be evaluated in this study employing realist evaluation methodology. Realist evaluation address "what works, for whom, in which contexts particular programmes do and don't work and what mechanisms are triggered by what programmes in what contexts" (27). Realist evaluation is useful to understand the interaction between context and mechanism in the intervention (27), to achieve the intended outcome of the HANDY program v. 2.0.

Context - Mechanism - Outcome Strategies identified in group-based peer-exchange activities targeting participants' ADL problems - ensures that participants experience a clear relationship between the first individual session and the group-based peer-exchange sessions - supporting motivation to participate in the group sessions targeting improvement of ADL ability

Engaging in the group-based peer-learning activity addressing reasons for ADL problems - expand the participants' understanding of their ADL problems, with a transactional perspective and not only related to hand function - supporting motivation for using compensatory strategies to improved ADL ability

Doing homework between sessions - make sense to the participants - supporting implementation of compensatory strategies at home to improved ADL ability

Study procedures Sample size The group-based occupational therapy program will be offered once in each municipality for eight participants. Accordingly, 2 x 16 participants with HOA will be recruited. This number of participants was determined based on a sample size large enough to provide information in relation to exploring mechanisms of action and evaluating trial design to determine if it is possible to proceed to a full scale RCT study (28,29).

Randomisation When baseline evaluations have been completed for 16 participants in a municipality, they will be randomised to either the HANDY occupational therapy intervention or a waiting list according to a computerized randomisation list. The randomisation process will be monitored including reasons to withdraw.

Data collection Data will be collected specifically to address each of the study aims. Moreover, participant demographic data will be collected. Participants with HOA and OTs will fill in registration forms independently.

Trial design, conduct and processes remaining feasibility aspects

Data collection methods

* Registration of participants handled by the OTs in each municipality.
* Registration forms filled in by participants with HOA following baseline, randomisation, and post intervention assessments.
* Diary entries filled in by participants with HOA.
* Completion rates of outcome measurements at baseline and post intervention. - Registration forms filled in by participants with HOA after each session.
* Semi-structured interviews with participants with HOA

Recruitment and retention To assess effectiveness of recruitment, randomisation and retention, the number of persons with HOA referred, and included in the pilot study, baseline and post-tests, the number and types of sessions received by the participants in the intervention group will be recorded consecutively by the OTs in each municipality. Furthermore, registration of participants randomised for the control group and their retention will also be registered at baseline and post-test.

Acceptability of trial in practice To evaluate acceptability of trial procedures in relation to progression criteria, this including randomisation and outcomes assessment procedures, participants with HOA will fill in registration forms addressing trial procedures following randomisation, baseline, and post intervention outcomes assessments. Ordinal response scales will be applied.

In a later full-scale RCT the outcome assessments will be as followed: Co-primary outcomes will be self-reported and observed ADL motor ability, and secondary outcomes will be observed ADL process ability, using the Activities of Daily Living Interview (ADL-I) (23) and Assessment of Motor and Process Skills (AMPS) (25,30), respectively. These instruments have previously been successfully applied in studies involving people with HOA, including the HANDY feasibility study (19).

Exploratory outcomes will in accordance with the Outcome Measures in Rheumatology (OMERACT) (30) be: Health-related quality of life (European Quality of life 5 Dimensions (EQ-5D)) (31); pain, stiffness and physical function (Australian Canadian Osteoarthritis Hand Index (AUSCAN) questionnaire (32); Patient global assessment (Visual Analogue Scale 0 to 100 mm) (33); and grip strength (GRIPPIT dynamometer)(34). These instruments are recommended and commonly used for people with HOA as in the COLOR trial (35). Further, exploratory outcomes in relation to goal attainment for participants will be evaluated with Goal Attainment Scale (GAS) (26). In the feasibility study GAS successfully captured changes of the participants goal attainment (19).

Breadth and selection of outcomes Based on results from the feasibility study, it was decided also to add a three-day dairy logbook as an exploratory outcome to assess real time activity level, occupational patterns and pain at baseline and post intervention outcomes assessments. More specifically, the time-geographic method will be used (36,37). The appropriateness of this outcomes will be evaluated based on the extent to which diary entries are filled in by participants with HOA. Additionally, if overall description of the participants real time activity, occupation patterns and pain are possible.

Completion of measures The outcomes (ADL-I, AMPS, GAS, EQ-5D, AUSCAN, Patient global assessment (VAS) and GRIPPIT) will be evaluated in relation to completion rates at baseline and post intervention.

Mechanisms of actions To explore the three specific topics in the preliminary program theory of the HANDY occupational therapy intervention (figure 2), participants with HOA will complete registration forms after each group session. Questions will address if the HANDY intervention supports improvement of identified ADL problems. Ordinal response scales will be applied.

Qualitative semi-structured interviews will be conducted with participants with HOA. This to explore the interaction between context and mechanism in the intervention, to achieve the intended outcome for the HANDY occupational therapy intervention. Interviews will be conducted in face-to-face focus groups corresponding with the occupational therapy intervention groups, immediately after completing the last session. Interviews will be carried out by two experienced researchers.

Feasibility and acceptability of intervention in practice To explore if the HANDY occupational therapy intervention v. 2.0 is feasible and acceptable, OTs and participants with HOA will fill out registration forms after each occupational therapy session (week 1-6). Questions in the registration forms will be a replication of questions asked in the feasibility study of the HANDY program v1.0, to determine if feasibility and acceptability have improved. Questions in the registration forms will address content and delivery of the components in each session of HANDY occupational therapy intervention v. 2.0. Ordinal response scales will be applied.

Progression criteria To determine if a full scale RCT can be recommended, progression criteria will be evaluated.

Data handling To ensure confidentiality, participants with HOA will hand in registration forms to the OT in closed envelopes at the end of each session. Data will be entered in a secure database.

Data analyses Nominal data will be reported based on numbers and percentages. Ordinal data and continuous data with lack of normal distribution will be presented based on medians and ranges. Participant demographic data will be presented, for participants with HOA (age, sex, social status and level of education) for OTs (age, sex and years of education).

Data related to the effectiveness of recruitment, randomisation and retention, and also completion of outcome measures, will be presented in a flow chart. Registration forms on acceptability of study procedures will include responses "yes/no" and Likert scales (from 1=to a very low degree to 5=to a very high degree), with the possibility of adding comments. in These data will be presented with median and range. Data on the appropriateness of outcomes and measurements, or more specifically on the three-day diary logbook, will be evaluated in relation to the extent of completion of diary entries.

To explore preliminary mechanisms of actions, data in registration forms, asking 'if identified ADL task performance problems were addressed in the group sessions', were based on Likert scales (from 1=to a very low degree to 5=to a very high degree). These data will be presented with median and range. Moreover, interview data will be transcribed verbatim and read through to get a sense of the whole. Hereafter, in relation to the three specific topics of the preliminary program theory, units will be identified and within each unit meaning units will be condensed.

Finally, to explore if the revised HANDY program (v 2.0) is feasible and acceptable, based on adjustments made, data from registration forms ("yes/no" and Likert scales (from 1=to a very low degree to 5=to a very high degree)) will be analyzed and compared with the result from the feasibility study of HANDY program (v 1.0) to explore if the program has been improved. To analyse if a full scale RCT can be recommended, progression criteria has been developed based on recommendation by Mellor et al (38).

Ethical The study will be conducted in accordance with the Helsinki declaration and Danish law. Informed consent will be obtained from each participant, including people with HOA and OTs, emphasizing the right to withdraw from the study at any time. A copy of the consent form will be provided to participants and the first author will be responsible for saving a consent form in the participant's study file. Each participant is given an ID number, with which all data is pseudonymized and only accessed by authorized personnel obliged to secrecy.

To minimize any risk all OTs will receive training in the procedures of the HANDY program and the delivery will be done by educated and experienced personal. The results of the study will be reported in accessible formats to study participants, decision makers in the participating municipalities, other stakeholders involved in the study, and public in general. Further, results will be published in peer-reviewed journals and presented on national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed by general practitioner with hand osteoarthritis
* Aged > 18 years
* Experiencing decreased ADL ability

Exclusion Criteria:

* Severe vision loss
* Severe hearing loss
* Cognitive deficits affecting the ability to engage in peer-learning activities
* Unable to participate in two or more group sessions due to other scheduled activities (e.g. holidays/travels).
* Acute illness is the primary reason for decreased ADL ability (Will be referred to other services in the municipality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Observed ADL motor ability | up to 3 months
  Change in observed ADL motor ability, using the Assessment of Motor and Process Skills (AMPS). Raw ordinal scores are converted into linear, interval scale (i.e. infinite scale) measures of ADL motor ability based on Rasch measurement models and reported in logits. Higher measures indicate higher ADL motor ability
Selfreported ADL ability | up to 3 months
  Change in self-reported ADL ability, using the standardised ADL-Interview (ADL-I). Raw ordinal scores are converted into linear, interval scale (i.e. infinite scale) measures of self-reported ADL ability based on Rasch measurement models and reported in logits. Higher measures indicate higher self-reported ADL ability

SECONDARY OUTCOMES:
Observed ADL process ability | up to 3 months
  Change in observed ADL motor ability, using the Assessment of Motor and Process Skills (AMPS). Raw ordinal scores are converted into linear, interval scale (i.e. infinite scale) measures of ADL process ability based on Rasch measurement models and reported in logits. Higher measures indicate higher ADL process ability

OTHER OUTCOMES:
Selfreported health-related quality of life | up to 3 months
  Selfreported health-related quality of life will be assessed by the European Quality of life 5 Dimensions (EQ-5D) including five quistions and visual analogue scale. The five quistions (Mobility; Self-care; Usual activities; Pain/Discomfort; Anixiety/Depression) on a likert scale 1 to 5 (1= very low degree, 5= very high degree). The visual analogue scale (0 to 100) with zero representing the worst health imagined and 100 the best health imagined.
Selfreported pain | up to 3 months
  Change in selfreported hand pain will be assessed using the Australian Canadian Osteoarthritis Hand Index (AUSCAN) questionnaire . AUSCAN items are rated on a visual analogue scale from zero mm (no symptoms) to 100 mm (worst symptoms), AUSCAN pain subscales will be reported in cm based on item sum scores for each subscale: pain (five items, score 0 to 50).
Selfreported stiffness | up to 3 months
  Change in selfreported hand stiffness will be assessed using the Australian Canadian Osteoarthritis Hand Index (AUSCAN) questionnaire. AUSCAN items are rated on a visual analogue scale from zero mm (no symptoms) to 100 mm (worst symptoms), AUSCAN subscales were reported in cm based on item sum scores for each subscale: stiffness (one item, score 0 to10).
Selfreported function | up to 3 months
  Selfreported function function will be assessed using the Australian Canadian Osteoarthritis Hand Index (AUSCAN) questionnaire. AUSCAN items are rated on a visual analogue scale from zero mm (no symptoms) to 100 mm (worst symptoms), AUSCAN subscales were reported in cm based on item sum scores for each subscale: function (nine items, score 0 to 90).
Patient global assessment | up to 3 months
  Patient global assessment will be measured on a Visual analogue scale (0 to 100) with zero representing the worst health and 100 the best health.
Grip strength | up to 3 months
  Change in grip strength will be measured in Newton (N) with the dynamometer GRIPPIT
Goal achievement | up to 2 months
  Goal achievement will be measured using the Goal Attainment Scale. The person with HOA and the OT will collaborate to formulate goals for the intervention and rated on a scale from -2 to +2, higher number indicates goal achivement.
Dairy logbook | up to 3 months
  A three-day dairy logbook as an exploratory outcome to assess real time activity level, occupational patterns and pain at baseline and post intervention. More specifically, the time-geographic method will be used.
Registation forms from people with hand osteoarthritis | up to 2 months
  Registration forms from people with hand osteoarthritis concerning perception of content and delivery in relation to HANDY program version 2.0. Registration forms designed for the study concern: 1) Likert scale 1 to 5 (1= very low degree, 5= very high degree). Questions to people with hand osteoarthritis in relation to the perception of content in GP and OT sessions.
Registration forms from Occupational therapist | up to 2 months
  Registration forms designed for the study concern: 1) Yes/NO questions in rela-tion to whether the instructions for occupational intervention session were followed. If No the OT can ad a comment about reason and how deviation was made 2) Likert scale 1 to 5 (1= very low degree, 5= very high degree). Questions in relation to the relevance of content in the occupational intervention session

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
If a data transfer is requested, the Capital Region of Denmark's legal department will decide in specific cases whether this is possible.

REFERENCES:
- [Background] Mellor K, Albury C, Dutton SJ, Eldridge S, Hopewell S. Recommendations for progression criteria during external randomised pilot trial design, conduct, analysis and reporting. Pilot Feasibility Stud. 2023 Apr 15;9(1):59. doi: 10.1186/s40814-023-01291-5. PMID 37061720
- [Background] Wallstrom A, Nordenskiold U. Assessing hand grip endurance with repetitive maximal isometric contractions. J Hand Ther. 2001 Oct-Dec;14(4):279-85. doi: 10.1016/s0894-1130(01)80006-5. PMID 11762728
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Wittrup-Jensen KU, Lauridsen J, Gudex C, Pedersen KM. Generation of a Danish TTO value set for EQ-5D health states. Scand J Public Health. 2009 Jul;37(5):459-66. doi: 10.1177/1403494809105287. Epub 2009 May 1. PMID 19411320
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Wong G, Westhorp G, Manzano A, Greenhalgh J, Jagosh J, Greenhalgh T. RAMESES II reporting standards for realist evaluations. BMC Med. 2016 Jun 24;14(1):96. doi: 10.1186/s12916-016-0643-1. PMID 27342217
- [Background] von Bulow C, Waehrens EE, Andersen U, Amris K, la Cour K. How a group-based occupational therapy program works in woman with fibromyalgia: A process evaluation of the ADAPT program. Scand J Occup Ther. 2023 Nov;30(8):1523-1540. doi: 10.1080/11038128.2023.2242380. Epub 2023 Aug 9. PMID 37557901
- [Background] Hansen AO, Kristensen HK, Cederlund R, Moller S, Tromborg H. An occupation-based intervention in patients with hand-related disorders grouped using the sense of coherence scale-A randomized controlled trial. J Hand Ther. 2020 Oct-Dec;33(4):455-469. doi: 10.1016/j.jht.2019.12.009. Epub 2020 Mar 7. PMID 32156580
- [Background] Hand C, Law M, McColl MA. Occupational therapy interventions for chronic diseases: a scoping review. Am J Occup Ther. 2011 Jul-Aug;65(4):428-36. doi: 10.5014/ajot.2011.002071. PMID 21834458
- [Background] Steultjens EM, Dekker J, Bouter LM, Leemrijse CJ, van den Ende CH. Evidence of the efficacy of occupational therapy in different conditions: an overview of systematic reviews. Clin Rehabil. 2005 May;19(3):247-54. doi: 10.1191/0269215505cr870oa. PMID 15859525
- See also: Related Info — https://www.frederiksberghospital.dk/afdelinger-og-klinikker/parker-instituttet/forskning/forskning-i-afdelingen/Sider/HANDY-projektet.aspx